CLINICAL TRIAL: NCT00743704
Title: Novel Noninvasive Techniques to Study Neutrophil Airway Inflammation in an Ozone Challenge Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Jens Hohlfeld, MD, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 08/04 Ozelot
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Other: ozoneexposure — subjects will be exposed to either ozone (250 ppb) or filtered air in an ozone challenge chamber for three hours. Ventilation will be increased to 20 l/min/m2 by intermittent exercise on a bicycle ergometer.

SUMMARY:
The primary objective of this pilot study is to establish a model of neutrophil airway inflammation for future testing of anti-inflammatory substances in an early stage of clinical development. Moreover, the suitability of an electronic nose for early detection and diagnosis of airway inflammation will be determined.

DETAILED DESCRIPTION:
Experimental ozone exposure of human subjects is known to induce transient neutrophilic airway inflammation with sputum neutrophilia and elevated concentrations of inflammatory mediators in bronchoalveolar lavage and sputum supernatants. In this study, ozone at a concentration of 250 ppb will be inhaled for three hours in an ozone challenge chamber.

In a recent study, ozone challenge has been discussed as a model for pulmonary diseases dominated by neutrophilic inflammation such as COPD, providing the possibility to test new anti-inflammatory substances in early stages of clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Healthy male and female nonsmokers, aged 18 to 55 years, with a history of less than 1 packyear having been nonsmokers for at least the last five years, FEV1 ≥ 80 % of predicted, FEV1/FVC ≥ 70 %
* Available to complete all study measurements
* Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by pregnancy test, and not nursing
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit)
  * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study -, implants, injectables, combined oral contraceptives, hormonal IUDs)
* Subjects must be able to produce adequate sputum
* Subjects must be responsive to ozone in a screening challenge (250 ppb, 3h) defined by a ≥ 10 % increase in sputum neutrophils 6 h after the start of ozone exposure

Exclusion Criteria:

* Upper or lower respiratory tract infection in the last four weeks prior to screening
* Subjects with a positive skin prick test to common aeroallergens will be excluded
* Past or present disease, which as judged by the investigator, may affect the outcome of the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
* Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
* Participation in another clinical trial 30 days prior to enrolment
* Administration of corticosteroids within the last 4 weeks prior to screening
* History of drug or alcohol abuse
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change of smellprints in exhaled breath | at the end of ozone exposure and 6 h and 24 h after the start of challenge compared with baseline and exposure to filtered air

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer-Institut für Toxikologie und Experimentelle Medizin, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Biller H, Holz O, Windt H, Koch W, Muller M, Jorres RA, Krug N, Hohlfeld JM. Breath profiles by electronic nose correlate with systemic markers but not ozone response. Respir Med. 2011 Sep;105(9):1352-63. doi: 10.1016/j.rmed.2011.03.002. Epub 2011 Mar 24. PMID 21439804